CLINICAL TRIAL: NCT02914145
Title: Mass Drug Administration of Monthly DHA-PQP to Accelerate Towards Malaria Elimination in Magude District, Southern Mozambique
Brief Title: Mass Drug Administrations of DHA-PQP to Accelerate Towards Malaria Elimination in Magude District, Southern Mozambique
Acronym: MDAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201/CNBS/15
Record Dates: First submitted 2016-09-14; First posted 2016-09-26 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants (Other): Any individual from the study area who participates and is medicated with DHAp in the mass drug administration campaign
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — Mass drug administration
  Other Names: Eurartesim

SUMMARY:
In line with the global and regional efforts towards malaria elimination, a five year program was established to assist the NMCP in adopting targeted evidence-based elimination plans through a 'learn by doing' strategy. The project aims to generate knowledge as data is generated to inform the programmatic aspects of the elimination plan, most importantly how to clear malaria parasites from the asymptomatic reservoir.

DETAILED DESCRIPTION:
This study aims to deliver two yearly consecutive rounds of community wide MDA using DHA-PQP (full treatment, 3 days, only supervised as DOT on day 0) at months 1 and 2, combined with parasite prevalence surveys using RDTs and PCR.

The first RDT survey (conducted to the entire study population of 60,000 inhabitants before each individual's dose of MDA1) would provide a precise estimate of RDT measurable P. falciparum baseline prevalence. During this first round of MDA, full blood will also be collected in filter papers for all individuals for PCR evaluation to investigate PCR-based parasite prevalence in the community. During the second MDA round, blood will be collected in filter papers in a subsample of the study population for screening of PCR-based parasite prevalence in the community and among first-trimester pregnant women.

Effectiveness of the MDA rounds will be measured throughout a 12-month period.

During the first six months, impact will be measured based on RDT positivity and PCR positivity measured on month 1 (baseline; both methods) and subsequently (month 2, only PCR; month 6, both RDT and PCR); and on malaria incidence in the community measured through passive case detection (PCD) in the different health posts. The success of the two rounds of MDA, as measured by: a) Prevalence of malaria infection (by RDT and/or PCR) in a subgroup of the study population on month six; b) Incidence of malaria as detected through PCD (from months 1 to 6); c) Identification of hotspots of maintained transmission in the study area; or d) Coverage achieved of MDA1 and MDA2 rounds). Should the two rounds not achieve the predefined success milestones [1. Decrease in parasite prevalence by 90% by RDT and/or PCR; 2) Coverage of 80% or above for both rounds; 3) Absence of clear geographic hotspots and 4) Incidence of clinical malaria in the community<1% i.e <600 cases/year] a two more round of MDA (or a more targeted focal MDA) in the totality or a part of Magude district will be organized, starting on month 7.

DHA/PQP has been chosen as the drug of choice for MDA. The pharmacokinetic profile of piperaquine - the long half-life component drug in DHA-PQP - confers a minimum of a 1-month post-treatment prophylaxis effect. If administered monthly (for 3 days at a time) with a 4 weeks interval, the prophylactic effect could protect individuals from pre-treatment Plasmodium infected mosquitoes as well as from mosquitoes infected after mass treatment from residual circulating gametocytes. Mosquitoes live for a maximum of 28 days during which they return to feed from humans. During this period the population of pre-treatment infected mosquitoes will gradually die away, exhausting the mosquito reservoir of infection.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who consent to participate in the study
* Residents in the study area
* Older than 6 months of age (or weighing more than 5Kg)
* Women in the second or third trimester who are not on IPTp

Exclusion Criteria:

* Individuals who do not consent to participate in the study
* Younger than 6 months of age (or weighing more than 5Kg)
* Women in the first trimester of pregnancy
* Severely ill individuals
* Individuals on contra-indicated medication

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240502 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Decrease in Parasite prevalence according to RDT | 6 months
  the proportion of individuals (according to age group) with P. falciparum infection (detected by RDT) out of all tested individuals (in that age group)
Decrease in Parasite prevalence according to PCR | 6 months
  as the proportion of individuals (according to age group) with P. falciparum infection (detected by PCR) out of all tested individuals (in that age group)
Total and confirmed outpatient (OPD) malaria case incidence and inpatient (IPD) malaria case incidence among all ages | 12 months
  the number of OPD and IPD malaria parasitologically confirmed cases per person per year, as ascertained from the routine passive case detection system utilizing facility catchment population size estimates as denominator.

SECONDARY OUTCOMES:
Population coverage of the MDA intervention | 3 weeks
  the proportion of individuals (≥6 months old) that agreed to participate in the MDA intervention and took under DOT the first dose of the 3-day long treatment of DHA-PQP among all individuals ≥6 months old eligible to participate in the intervention in the target population.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Aide, MD, MSc, PhD, Study Director — pedro.aide@manhica.net

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740
- [Derived] Thomas R, Cirera L, Brew J, Saute F, Sicuri E. The short-term impact of a malaria elimination initiative in Southern Mozambique: Application of the synthetic control method to routine surveillance data. Health Econ. 2021 Sep;30(9):2168-2184. doi: 10.1002/hec.4367. Epub 2021 Jun 8. PMID 34105200
- [Derived] Galatas B, Saute F, Marti-Soler H, Guinovart C, Nhamussua L, Simone W, Munguambe H, Hamido C, Montana J, Muguande O, Maartens F, Luis F, Paaijmans K, Mayor A, Bassat Q, Menendez C, Macete E, Rabinovich R, Alonso PL, Candrinho B, Aide P. A multiphase program for malaria elimination in southern Mozambique (the Magude project): A before-after study. PLoS Med. 2020 Aug 14;17(8):e1003227. doi: 10.1371/journal.pmed.1003227. eCollection 2020 Aug. PMID 32797101
- [Derived] Galatas B, Nhacolo A, Marti H, Munguambe H, Jamise E, Guinovart C, Cirera L, Amone F, Macete E, Bassat Q, Rabinovich R, Alonso P, Aide P, Saute F, Sacoor C. Demographic and health community-based surveys to inform a malaria elimination project in Magude district, southern Mozambique. BMJ Open. 2020 May 5;10(5):e033985. doi: 10.1136/bmjopen-2019-033985. PMID 32371510